CLINICAL TRIAL: NCT06936358
Title: Comparison of the Effect of Injectable Platelet-rich Fibrin and Advanced Platelet-rich Fibrin With Xenograft on the Socket Preservation of Mandibular Extracted Molars ( a Randomised Controlled Clinical Trial) Comparison of the Effect of Injectable Platelet-rich Fibrin and Advanced Platelet-rich Fibrin With Xenograft on the Socket Preservation of Mandibular Extracted Molars ( a Randomised Controlled Clinical Trial)
Brief Title: Injectable Platelet-rich Fibrin and Advanced Platelet-rich Fibrin With Xenograft on the Socket Preservation of Mandibular Extracted Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0663_04/2023
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Tooth Extraction; Socket Preservation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator)
  Interventions: Other: Control
- A-PRF (Experimental)
  Interventions: Other: A-PRF
- I-PRF (Experimental)
  Interventions: Other: I-PRF

INTERVENTIONS:
Other: Control — Control group received bone graft alone after extraction
  Arms: Control
Other: A-PRF — 30 mL of whole venous blood will be withdrawn from the antecubital vein via scalp vein catheter centrifuged at 1500 rpm for 14 minutes.
  Arms: A-PRF
Other: I-PRF — 30 mL of whole venous blood will be withdrawn from the antecubital vein via scalp vein catheter centrifuged at 700 rpm for 3 minutes
  Arms: I-PRF

SUMMARY:
Different materials and techniques are employed for socket preservation to reduce the alveolar bone resorption in both the horizontal and vertical dimensions as well as the soft tissue collapse after tooth extraction. Because of the repair abilities of the growth factors and proteins released by platelets, the development and application of platelet-enriched preparations have revolutionised the area of regenerative medicine.The present study will be designed to study the difference between A-PRF and IPRF with the addition of Xenograft in the preservation of bone in mandibular molars.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need extraction of hopeless mandibular molars
* Teeth with advanced caries not amenable for conservative treatment
* Patients who are willing and fully capable of complying with the study protocol.

Exclusion Criteria:

* Systemic diseases that prevent surgery
* Acute or chronic oral infections
* Periodontal diseases
* Heavy smokers or alcoholics
* On anticoagulant drugs.
* Pregnancy
* History of radiotherapy or chemotherapy of the head and neck region

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Change in healing | Baseline and 12 weeks
  A modified Landry, Turnbull, and Howley healing index will be used to assess wound healing (HI). This entails evaluating the following parameters in a comparative manner using a dichotomic score (1/0). Tissue colour or the presence or absence of redness to indicate inflammatory processes; granulation tissue; suppuration; swelling; degree of tissue epithelialisation (partial or complete); and the presence or absence of bleeding and tenderness on palpation
change in bone density | Baseline and 12 weeks
  Bone density will be measured using CBCT examinations

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt